CLINICAL TRIAL: NCT05975866
Title: The Effects of an Anti-inflammatory Diet With or Without Curcumin Supplementation on Anthropometric Measurements, Concentrations of Thyroid Hormones, Anti-TPO, and Systemic Inflammation in Plasma and NFK-B in Peripheral Blood Mononuclear Cells in Patients With Hashimato
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, MD-PHD of nutrition s science, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0410359181
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Thyroid Diseases; Hypothyroidism; Hashimoto Disease
Keywords: Thyroid Diseases; Hypothyroidism; Hashimoto Disease; Anti-inflammatory diet; Curcumin
MeSH Terms: conditions — Thyroid Diseases; Hypothyroidism; Hashimoto Disease | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: The study subjects are Hashimoto's patients who, if they wish to participate in this research, a written consent form will be obtained from the patients at the beginning of the study. The patients will be classified according to age and sex. Then, using Stratified Block Randomization, patients will be placed in one of two intervention or placebo groups. The intervention will last 12 weeks, and the anti-inflammatory diet will be personalized based on each person's calorie intake. Patients will be asked to take one tablet with cold water daily (morning, noon, and night with the main meals). Also, the curcumin placebo in size, shape, color, appearance, smell, and dispensing cans of the drug will be similar to the curcumin supplement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the start of the study, the set of cans containing the relevant capsules will be coded as A and B by someone other than the researcher so that the researcher does not know the type of capsule received by the patients. The cans containing the relevant capsules will be delivered to the patients on a monthly basis, and they will be asked to take one tablet with cold water every day (morning, noon, and night with the main meals). Also, the curcumin placebo will be similar to the curcumin supplement in terms of size, shape, color, appearance, smell, and drug distribution cans.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group receiving anti-inflammatory diet with curcumin supplement (Experimental): Implementation of an anti-inflammatory diet along with the daily consumption of three 500 mg curcumin capsules along with the main meals of breakfast, lunch, and dinner.
  Interventions: Dietary Supplement: curcumin; Behavioral: Anti-inflammatory diet
- Group receiving anti-inflammatory regimen with curcumin placebo (Placebo Comparator): Implementation of an anti-inflammatory diet along with the daily consumption of three 500 mg placebo capsules of curcumin (microcrystalline cellulose) and the main meals of breakfast, lunch, and dinner.
  Interventions: Behavioral: Anti-inflammatory diet

INTERVENTIONS:
Dietary Supplement: curcumin — Daily consumption of three 500 mg curcumin capsules with breakfast, lunch, and dinner
  Arms: The group receiving anti-inflammatory diet with curcumin supplement
Behavioral: Anti-inflammatory diet — The anti-inflammatory diet will be personalized based on each person's calorie intake in five meals. Achieving the goals of an anti-inflammatory diet by consuming only one type of food or following its principles in one meal is impossible and must be implemented consistently and regularly in a meal plan.

SUMMARY:
The goal of this clinical trial is to investigate The effects of an anti-inflammatory diet with or without curcumin supplementation on anthropometric measurements, concentrations of thyroid hormones, anti-TPO, and systemic inflammation in plasma and NFK-B in peripheral blood mononuclear cells in patients with Hashimoto.

The main questions it aims to answer are:

1. Does prescribing an anti-inflammatory diet with or without curcumin supplementation significantly affect the changes in anthropometric measurements (weight, body mass index, BMI, waist circumference, waist-to-hip ratio) in patients with Hashimoto's disease?
2. Does prescribing an anti-inflammatory diet with or without curcumin supplementation significantly affect the changes in the serum concentration of thyroid hormones (T3, T4, TSH) in patients with Hashimoto's disease?
3. Does prescribing an anti-inflammatory diet with or without curcumin supplementation significantly affect the change of Anti-TPO concentration in patients with Hashimoto's disease?
4. Does prescribing an anti-inflammatory diet with or without curcumin supplementation significantly affect the changes in systemic inflammation indicators (hs-CRP, IL-6) in plasma and NF-κB in peripheral blood mononuclear cells in patients with Hashimoto's disease?

ELIGIBILITY:
Inclusion Criteria:

Having Hashimoto's thyroiditis Willingness to cooperate Body mass index between 35 and 18.5 TSH less than ten and without clinical symptoms Not taking levothyroxine tablets

Exclusion Criteria:

Pregnancy and breastfeeding kidney Diseases Follow non-routine weight loss diets for three months before the start of the study × Taking slimming and fat-burning drugs, fiber powder Mineral, vegetable, and fiber vitamin supplements

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-23 (Estimated); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
IL6 | 3 month
  Interleukin 6
hs-Crp | 3 month
  high-sensitivity C-reactive protein
NF-KB | 3 month
  Nuclear factor kappa-light-chain-enhancer of activated B cells
Anti-tpo | 3 month
  antithyroperoxidase
T4 | 3 month
  Thyroxine
T3 | 3 month
  Triiodothyronine
TSH | 3 month
  Thyroid-stimulating hormone
waist circumference | 3 month
  waist circumference in Centimeter
hip circumference | 3 month
  hip circumference in Centimeter
waist to hip ratio | 3 month
  an Anthropometric index
BMI | 3 month
  Body Mass Index - Anthropometric index
Total Cholestrol | 3 month
  serum lipid profile
TG | 3 month
  Triglyceride - serum lipid profile
Hb | 3 month
  hemoglobin - Blood test
hematocrit | 3 month
  Blood test
LDL | 3 month
  low-density lipoprotein
HDL | 3 month
  high-density lipoprotein

CONTACTS AND LOCATIONS:
Locations (1):
- Golbon Sohrab, Tehran, National Nutrition and Food Technology Research Institute, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourbour F, Mahdavi B, Naghshi N, Yari Z, Hosseini SM, Kalbasi S, Sohrab G. The Combined Effects of an Anti-Inflammatory Diet and Curcumin Supplementation on Thyroid Function and Lipid Profile in Patients With Hashimoto's Thyroiditis: A Double Blind Randomised Clinical Trial. Endocrinol Diabetes Metab. 2026 Jan;9(1):e70138. doi: 10.1002/edm2.70138. PMID 41329567